CLINICAL TRIAL: NCT06592885
Title: Evaluation of Success of Hall Technique Versus Atraumatic Restorative Treatment in the Management of Carious Primary Molars: a Randomized Clinical Trial
Brief Title: Comparing Minimally Invasive Techniques Used in Treatment of Carious Primary Molars in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Atef Ahmed, Principal invistigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HT Vs ART in pedodontics
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hall Technique in treatment of carious primary molars (Active Comparator): The Hall technique, proposed by Norna Hall in the 1980s, involves the placement of preformed metal crowns on primary molars without any tooth preparation or local anesthesia
  Interventions: Procedure: Hall Technique in treatment of carious primary molars
- Atraumatic Restorative Treatment in treatment of carious primary molars (Experimental): ART, which took place in Tanzania during the mid-1980s, is a conservative approach involving the removal of carious lesions using hand instruments, followed by the application of a glass ionomer restoration, promoting the preservation of tooth structure.
  Interventions: Procedure: Atraumatic Restorative Treatment in treatment of carious primary molars

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment in treatment of carious primary molars — ART, which took place in Tanzania during the mid-1980s, is a conservative approach involving the removal of carious lesions using hand instruments, followed by the application of a glass ionomer restoration. This technique aims to be minimally invasive, promoting the preservation of tooth structure. The ART technique, employed in situations where ideal clinical conditions are challenging to achieve, has demonstrated effectiveness as a reliable method for managing cases where conventional treatment methods face resistance from children . However, concerns exist regarding the longevity of ART restorations and the impact of operator skill on outcomes.
  Arms: Atraumatic Restorative Treatment in treatment of carious primary molars
Procedure: Hall Technique in treatment of carious primary molars — The Hall technique, proposed by Norna Hall in the 1980s, involves the placement of preformed metal crowns on primary molars without any tooth preparation or local anesthesia.
  Advocates of the Hall technique emphasize its simplicity, reduced need for traditional drilling, and high reported success rates in clinical studies.
  However, concerns have been raised regarding long-term aesthetics and potential psychological impacts due to the visibility of metal crowns.
  Arms: Hall Technique in treatment of carious primary molars

SUMMARY:
Dental caries is a natural process by which bacteria in the biofilm causes fluctuations in the pH, which leads to enamel erosion and result in visible lesions. If left untreated, caries will progress and result in pain, abscess, and systemic infection, leading to functional and/or psychosocial impairment which is a serious problem Caries is, in fact, the most prevalent childhood disease in the world and is most prominent among low-economic populations. So, the main goal is to minimize Dental caries as much as possible by applying preventive measures to reduce the occurrence and progression of dental caries.

In that scope, both Atraumatic Restorative Treatment (ART) and the Hall Technique (HT) were created as part of Minimal Invasive Dentistry (MID) to slow the downward restorative spiral and reduce discomfort during the treatment as neither of which requires the administration of local anesthesia nor the use of rotary instruments.

According to a retrospective analysis, utilizing the Hall technique to seal cavities performed much better than using conventional restorations. statistically and clinically during 10 years of follow-up.

Since ART is associated with lower levels of anxiety, pain, and discomfort than traditional dentistry procedures, it has become widely employed in pediatric dentistry. Despite having reduced survival rates in multiple-surface restorations, ART is still regarded as a viable, evidence-based choice for treating and preventing caries lesions in primary posterior teeth since it is a quick, inexpensive, and comfortable procedure for the patient.

DETAILED DESCRIPTION:
One of the most prevalent childhood diseases, dental caries, affects up to 90% of children globally, especially those from the underprivileged group.

WHO estimates that Egypt has a 60% prevalence of dental caries. Early childhood caries has a negative effect on a child's oral health-related quality of life. Both the family and the child are directly affected.

The ideal treatment of carious lesions has been the subject of recent revolutions. Traditional restorative methods, which focused on completely removing carious tooth tissue and then placing a restoration have been replaced by more biological and minimally invasive methods that concentrate on controlling biofilms and disrupting the cariogenic biofilm environment to stop caries.

The Hall Technique (HT) supports this theory. Without any dental preparation or caries removal, a preformed metal crown (PMC) is simply fixed to the carious tooth using glass ionomer cement (GIC). The cariogenic biofilm beneath the cap is sealed.

The Hall technique of stainless- steel crown placement has proved to be a viable restorative option for carious primary molars resulting in its successful exfoliation.

Management techniques would include atraumatic restorative treatment as well as those in which dentine carious tissue is selectively removed to soft or firm dentine in a single session (ART).

ART has been widely used in pediatric dentistry because it is linked with lower levels of anxiety, pain, and discomfort, as well as better acceptance by children, compared to conventional treatment.

ART uses only hand instruments to remove carious tissue and prepare the cavity. Additional extended clinical investigations are required to assess the effectiveness of these methods in addressing carious lesions on diverse tooth surfaces and various dentin layers and to provide evidence supporting the integration of these techniques into standard practice.

Since there is a need for further research, with larger sample sizes and extended follow-up durations in Egypt, to assess the effectiveness of these methods for treating carious primary teeth, this study will be conducted.

This research aims to compare the success of the Hall Technique to the Atraumatic Restorative treatment in the management of carious primary molars in children.

ELIGIBILITY:
Inclusion Criteria:

1. Age: From 4 to 6 years.
2. Caries in primary molars within enamel/dentin with vital pulp.
3. Healthy children.
4. Cooperative children.

Exclusion Criteria:

1. Presence of signs and symptoms of necrosis.
2. Root caries.
3. History of Spontaneous pain.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Success, Assessed by clinical examination | From enrollment to the end of treatment at 12 months (with follow up at 3-6-9-12 months)
  * Standard clinical criteria will be used to determine whether a restoration (ART/HT) was successful or not in terms of having a satisfactory restoration that requires no further intervention and also the absence of any signs or symptoms of pulp damage.
  * Measuring unit is Binary (Yes/No)

SECONDARY OUTCOMES:
Post-operative pain and discomfort | Measured immediately after placement of SSC or restoration
  Immediately after the treatment, any pain and discomfort experienced by the child will be recorded using the Face Pain Scale - revised (FPS-R), which has six numbered faces from 0 to10. Each child will be asked to mark the face that reflects her or his experienced pain during the treatment. There is no pain visible on the first face [indicating the face on the far left]. As you move from left to right, the faces get progressively more painful until you reach the last, which is incredibly painful [indicating the face on the far right]. The (FPS-R) faces will be scored as 0-2-4-6-8-10.
Child Behavior | Measured immediately after placement of SSC or restoration
  Venham Anxiety Rating Scale is a reliable system for rating behavior of children in the dental setting, a child's fear and lack of cooperation are assessed using five behaviorally defined categories, ranging from zero to five (Six-point scales 0-1- 2-3-4-5), which are included in each measure; higher values denote greater anxiety or an uncooperative manner.
Child Anxiety | Measured immediately after placement of SSC or restoration
  Venham behavior rating scale is a reliable system for rating the behavior of children in the dental setting.a child's fear and lack of cooperation are assessed using five behaviorally defined categories, ranging from zero to five (Six-point scales 0-1- 2-3-4-5), which are included in each measure; higher values denote greater anxiety or an uncooperative manner.
Canine overbite: HT | Measured in millimeters immediately after placement of pre-fabricated stainless steel crown (SSC)
  1. The canine overbite will be calculated in millimeters before the preparation by measuring the distance between the incisal points of the maxillary canine on the same side of the mouth to the gingival zenith of the mandibular canine using a Boley's Gauge.
  2. If checking the same side was not possible (e.g., loss of canine) the distance between canines on the other side will be measured.
  3. These prefabricated SSCs will be pre-trimmed to the optimum length, belled, and pre-crimped at the cervical margin.
  4. The SSC will be loaded with glass ionomer luting cement and partially fitted on the tooth using a finger. The patient will be asked to bite on a cotton roll and the SSC will be fully seated.
  5. Excess cement will be removed; Post-treatment overbite (immediately after the treatment) will be recorded.
  6. Changes in the canine overbite will be determined by subtracting the follow-up canine overbite from the baseline (pretreatment).

CONTACTS AND LOCATIONS:
Overall Officials: Gihan Abou Elneil Professor of Pediatric Dentistry and Dental Public Health, Professor, Study Director — Cairo University; Ahmed El. Khadem Associate Professor of Pediatric Dentistry, Associate Professor, Study Director — Cairo University; Dr. Shereen Hassan El-Shamy Lecturer of Pediatric Dentistry, Study Director — Cairo University
Locations (1):
- Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kaptan A, Korkmaz E. Evaluation of success of stainless steel crowns placed using the hall technique in children with high caries risk: A randomized clinical trial. Niger J Clin Pract. 2021 Mar;24(3):425-434. doi: 10.4103/njcp.njcp_112_20. PMID 33723119
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33723119/